CLINICAL TRIAL: NCT00310544
Title: Multicenter, Single-blind, Randomized, Intraindividual Study of the Safety and Efficacy of Magnevist Gadopentetate Dimeglumine (Magnevist® Injection) at 0.1 and 0.2 mmol/kg for the Depiction of Delayed Enhancement in Patients With Documented Myocardial Infarction
Brief Title: Depiction of Delayed Enhancement in Patients With Documented Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 91230; DE-03899; 306947
Record Dates: First submitted 2006-03-31; First posted 2006-04-04 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Gadolinium DTPA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Experimental)
  Interventions: Drug: Magnevist (Gadopentetate dimeglumine, BAY86-4882)
- Arm 1 (Experimental)
  Interventions: Drug: Magnevist (Gadopentetate dimeglumine, BAY86-4882)

INTERVENTIONS:
Drug: Magnevist (Gadopentetate dimeglumine, BAY86-4882) — One intravenous injection per period. Period 1 and 2 are separated by 4 to 14 days.period1:Magnevist 0.1 mmol/kg body weightperiod 2: Magnevist 0.2 mmol/kg body weight
  Arms: Arm 1
Drug: Magnevist (Gadopentetate dimeglumine, BAY86-4882) — One intravenous injection per period. Period 1 and 2 are separated by 4 to 14 days.period 1: Magnevist 0.2 mmol/kg body weightperiod 2: Magnevist 0.1 mmol/kg body weight
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine the dose of drug which is most effective in the delineation of dead heart muscle.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 8 weeks post-documented myocardial infarction (heart attack)

Exclusion Criteria:

* History of radiation therapy to the chest
* Clinically unstable
* Any contraindication for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-03; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Quantitative measurement of the total area of delayed enhancement | 30 min post injection

SECONDARY OUTCOMES:
Quantitative measures of area of delayed enhancement and signal intensities | At 5, 10 and 20 minutes post injection
Semiquantitative measures of area of delayed enhancement | At 5, 10, 20 and 30 minutes post injection
Presence of delayed enhancement | At 5,10 and 20 minutes post injection
Wall motion endpoints | Pre-injection
Safety | From baseline to 24h follow-up of second imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- United States (6):
  - San Diego, California
  - Winston-Salem, North Carolina
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Pittsburgh, Pennsylvania
- Buenos Aires, Buenos Aires, Argentina